CLINICAL TRIAL: NCT04862377
Title: Efficacy and Safety of the Intratracheal Administration of Budesonide With Porcine Pulmonary Surfactant in Very Preterm Infants to Prevent Bronchopulmonary Dysplasia: Randomized Clinical Trial (BuS Trial)
Brief Title: Intratracheal Budesonide With Surfactant to Prevent Bronchopulmmonary Dysplasia.
Acronym: BuS
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Hospital Clinic of Barcelona (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: BuS2020
Record Dates: First submitted 2021-03-05; First posted 2021-04-28 (Actual); Last update posted 2021-09-13 (Actual); Status verified 2021-04

CONDITIONS: Bronchopulmonary Dysplasia; Respiratory Distress Syndrome in Premature Infant; Prematurity
Keywords: Bronchopulmonary dysplasia; Respiratory Distress Syndrome in premature infant; Prematurity; Lung injury; Poractant alfa; Pulmonary surfactant; Budesonide; Anti-inflammatory agents; Glucocorticoids; Lung ultrasound; IL-6
MeSH Terms: conditions — Bronchopulmonary Dysplasia; Premature Birth; Lung Injury | interventions — poractant alfa; Budesonide

STUDY DESIGN:
Intervention Model Description: This is a randomised trial. Infants who fit criteria for surfactante administration will be randomly assigned into 2 groups: "Standard treatment group" receiving only intratracheal surfactant, and "Interventional treatment group" receiving intratracheal surfactant combined with budesoinde.
  It will be a third group of patients ≤32 weeks ("Control group") who won´t fit criteria for surfactant administration.
Who Masked: Participant
Masking Description: When eligibility of an infant is confirmed, consent will be obtained. Infants candidates to surfactant administration will be randomly assigned to either receive surfactant with budesonide, or surfactant alone, using a web-based randomisation system with an allocation ratio of 1:1.
  Primary care provider in charge of the patient at the time of the enrolment will be responsible for the randomization, and for the preparation of the drug (surfactant alone, or surfactant with budesonide).
  Participants will be masked.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Standard treatment group (Active Comparator): Infants randomised to the "standard treatment" arm will receive intratracheal surfactant as per usual clinical indications of respiratory distress syndrome in these preterm infants.
  In that sense, and based in those clinical indications, we have developed a risk calculator for surfactant administration in preterm infants ≤32 weeks GA. We will use it to decide what patients will receive surfactant (calculator available on: https://1drv.ms/x/s!Arjkl83HIXSngP8TWh8O6oi6Ztdw3w?e=gNCMxP).
  Interventions: Drug: Poractant Alfa Intratracheal Suspension [Curosurf]
- Interventional treatment group (Experimental): Infants randomised to the "interventional treatment" arm will receive intratracheal surfactant mixed with budesonide. Indication of surfactant, as equal as for the "standard treatment" arm, will be decided using the calculator.
  Interventions: Drug: Poractant Alfa Intratracheal Suspension [Curosurf]; Drug: Budesonide 0.5 MG/ML
- Control group (No Intervention): Infants ≤32 weeks with no indications for surfactant administration. Their clinical management will be the usual in our neonatal unit.

INTERVENTIONS:
Drug: Poractant Alfa Intratracheal Suspension [Curosurf] — Poractant alfa (Curosurf®):
  First dose of treatment: 200mg/Kg. Further doses (up to a total maximum of 3 within first 48 hours of life): 100mg/Kg.
  Other Names: Curosurf®
  Arms: Interventional treatment group; Standard treatment group
Drug: Budesonide 0.5 MG/ML — Poractant alfa (Curosurf®) + Budesonide nebulizer solution (Budesonida Aldo-Unión 0.5mg/mL suspensión para inhalación por nebulizador®):
  First dose: 200mg/Kg of surfactant + 0.25mg/Kg of budesonide. Further doses (up to a total maximum of 3 within first 48 hours of life): 100mg/Kg of surfactant + 0.25mg/Kg of budesonide.
  Other Names: Budesonida Aldo-Unión 0.5mg/mL suspensión para inhalación por nebulizador®
  Arms: Interventional treatment group

SUMMARY:
This study is designed to determine whether intratracheal administration of budesonide combined with surfactant, as compared to surfactant alone, will modify ecographic (lung ultrasound score) and biological markers (IL-6 concentration in respiratory secretions) at 7 days of life in preterm infants ≤32 weeks of gestational age (GA).

DETAILED DESCRIPTION:
Bronchopulmonary dysplasia (BPD) is one of the main morbidities associated with extreme prematurity and, despite the improvement of respiratory care in the latest years, overall incidence is not decreasing. Etiology of BPD is multifactorial and local inflammation plays an important role in it, therfore, local anti-inflammatory drugs could be effective in preventing BPD.

Recent randomised trials have shown a lower incidence of BPD/death with the use of a combination of budesonide with surfactat compared to surfactant alone, and further clinical trials are currently ongoing.

This is a controlled phase IV, randomised, unicenter clinical trial designed to evaluate the effect of intratracheal administration of budesonide combined with surfactant, as compared to surfactant alone, in BPD in preterm infants ≤32 weeks of GA. Investigators will compare ecographic and biological markers, as well as respiratory outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Infants born equal or earlier than 32 weeks of gestational age admitted in the Neonatal Intensive Care Unit.
* Parental consent signed.
* Less than or equal to 48 hours postnatal age.

Exclusion Criteria:

* Infants with known major congenital anomalies (eg. congenital upper airwayobstruction, congenital lung anomaly, severe pulmonary hypoplasia, hydrops,neuromuscular diseases, chromosomopaties)
* Infants with poor prognosis and risk of imminent death
* Infants who have received the first dose of surfactant before of the enrolment to the study.

Max Age: 48 Hours | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 50 (Estimated)
Dates: Start 2021-10-01 (Estimated); Primary Completion 2024-04-01 (Estimated); Study Completion 2026-04-01 (Estimated)

PRIMARY OUTCOMES:
Lung ultrasound score at 7 days of life. | 7 days of life
  LUS will be performed with the patients in supine position and slightly lying on the side of the taken view. Each lung will be divided in five areas through longitudinal orientation and images will be taken using the linear probe (VF 13-5MHz).
IL-6 concentration in respiratory secretions at 7 days of life. | 7 days of life
  Nasopharyngeal aspirate (NPA) will be collected by standard procedure. IL-6 concentration will be determined by Human IL-6 Quantikine ELISA (R&D Systems Inc., Minneapolis, MN, USA).

SECONDARY OUTCOMES:
Lung ultrasound score at 28 days of life. | 28 days of life
  LUS will be performed with the patients in supine position and slightly lying on the side of the taken view. Each lung will be divided in five areas through longitudinal orientation and images will be taken using the linear probe (VF 13-5MHz).
IL-6 concentration in respiratory secretions at 28 days of life. | 28 days of life
  Nasopharyngeal aspirate (NPA) will be collected by standard procedure. IL-6 concentration will be determined by Human IL-6 Quantikine ELISA (R&D Systems Inc., Minneapolis, MN, USA).
Number of days of oxygen | 7 and 28 days of age, 36 weeks of post-menstrual age.
  Number of days on FiO2 >21% supplied by any respiratory support
Number of days of respiratory support | 7 and 28 days of age, 36 weeks of post-menstrual age.
  Number of days on each level of respiratory support:
  * No respiratory support
  * Nasal cannula at flow rates ≤ 2L/min
  * Nasal cannula at flow rates > 2L/min
  * CPAP/BIPAP
  * Invasive mechanical ventilation
Mean airway pressure (MAP) | 7 and 28 days of age, 36 weeks of post-menstrual age.
  Maximum MAP mesured in cmH2O at 7 and 28 days of age, 36 weeks of postmenstrual age.
Incidence of bronchopulmonary dysplasia | 36 weeks of post-menstrual age.
  BPD will be defined according to the 2001 workshop definition (Jobe AH, Bancalari E. Bronchopulmonary dysplasia. American Journal of Respiratory and Critical Care Medicine. American Lung Association; 2001; pp 1723-9).
Respiratory status and neurodevelopment | 24 months of age.
  Neurodevelopment will be assessed using Bayley-III test.

CONTACTS AND LOCATIONS:
Overall Officials: Marta Teresa-Palacio, MD, Principal Investigator — Hospital Clinic of Barcelona

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Heo M, Jeon GW. Intratracheal administration of budesonide with surfactant in very low birth weight infants to prevent bronchopulmonary dysplasia. Turk J Pediatr. 2020;62(4):551-559. doi: 10.24953/turkjped.2020.04.004. PMID 32779407
- [Background] Oulego-Erroz I, Alonso-Quintela P, Terroba-Seara S, Jimenez-Gonzalez A, Rodriguez-Blanco S. Early assessment of lung aeration using an ultrasound score as a biomarker of developing bronchopulmonary dysplasia: a prospective observational study. J Perinatol. 2021 Jan;41(1):62-68. doi: 10.1038/s41372-020-0724-z. Epub 2020 Jul 14. PMID 32665687
- [Background] Alonso-Ojembarrena A, Lubian-Lopez SP. Lung ultrasound score as early predictor of bronchopulmonary dysplasia in very low birth weight infants. Pediatr Pulmonol. 2019 Sep;54(9):1404-1409. doi: 10.1002/ppul.24410. Epub 2019 Jun 10. PMID 31216121
- [Background] Forster K, Sass S, Ehrhardt H, Mous DS, Rottier RJ, Oak P, Schulze A, Flemmer AW, Gronbach J, Hubener C, Desai T, Eickelberg O, Theis FJ, Hilgendorff A. Early Identification of Bronchopulmonary Dysplasia Using Novel Biomarkers by Proteomic Screening. Am J Respir Crit Care Med. 2018 Apr 15;197(8):1076-1080. doi: 10.1164/rccm.201706-1218LE. No abstract available. PMID 29053024
- [Background] Venkataraman R, Kamaluddeen M, Hasan SU, Robertson HL, Lodha A. Intratracheal Administration of Budesonide-Surfactant in Prevention of Bronchopulmonary Dysplasia in Very Low Birth Weight Infants: A Systematic Review and Meta-Analysis. Pediatr Pulmonol. 2017 Jul;52(7):968-975. doi: 10.1002/ppul.23680. Epub 2017 Feb 6. PMID 28165675
- [Background] Yeh TF, Chen CM, Wu SY, Husan Z, Li TC, Hsieh WS, Tsai CH, Lin HC. Intratracheal Administration of Budesonide/Surfactant to Prevent Bronchopulmonary Dysplasia. Am J Respir Crit Care Med. 2016 Jan 1;193(1):86-95. doi: 10.1164/rccm.201505-0861OC. PMID 26351971
- [Background] Kuo HT, Lin HC, Tsai CH, Chouc IC, Yeh TF. A follow-up study of preterm infants given budesonide using surfactant as a vehicle to prevent chronic lung disease in preterm infants. J Pediatr. 2010 Apr;156(4):537-41. doi: 10.1016/j.jpeds.2009.10.049. Epub 2010 Feb 6. PMID 20138301
- [Background] Yeh TF, Lin HC, Chang CH, Wu TS, Su BH, Li TC, Pyati S, Tsai CH. Early intratracheal instillation of budesonide using surfactant as a vehicle to prevent chronic lung disease in preterm infants: a pilot study. Pediatrics. 2008 May;121(5):e1310-8. doi: 10.1542/peds.2007-1973. Epub 2008 Apr 21. PMID 18426851
- [Background] Aldecoa-Bilbao V, Balcells-Esponera C, Herranz Barbero A, Borras-Novell C, Izquierdo Renau M, Iriondo Sanz M, Salvia Roiges M. Lung ultrasound for early surfactant treatment: Development and validation of a predictive model. Pediatr Pulmonol. 2021 Feb;56(2):433-441. doi: 10.1002/ppul.25216. Epub 2020 Dec 23. PMID 33369257
- [Background] Jobe AH, Bancalari E. Bronchopulmonary dysplasia. Am J Respir Crit Care Med. 2001 Jun;163(7):1723-9. doi: 10.1164/ajrccm.163.7.2011060. No abstract available. PMID 11401896